CLINICAL TRIAL: NCT00773006
Title: Canadian Prospective, Observational Study on the Use of LMWH in the Setting of Percutaneous Coronary Intervention
Brief Title: Canadian Anticoagulant Percutaneous Coronary Intervention Registry
Acronym: CAPCIR
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Robert Welsh, Associate Professor, University of Alberta
Other Study IDs: CAPCIR02474
Record Dates: First submitted 2008-01-28; First posted 2008-10-16 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary intervention; anticoagulation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Stable/elective PCI patients
- B: NSTEMI PCI patients
- C: STEMI PCI patients

SUMMARY:
Advances in mechanical intervention (PCI) and anticoagulation therapy have been the cornerstone of treatment of patients with coronary artery disease. However, the large diversity of approaches to anticoagulation during PCI introduces gaps in knowledge regarding management of cardiac patients. As such, we have initiated a national PCI registry to elucidate anticoagulant choice, dosing strategies, case selection dynamics, and clinical outcomes in the Canadian health care environment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 or more years of age.
2. Undergoing PCI during treatment with LMWH
3. Provision of written and informed consent

Exclusion Criteria:

1. Language, medical, or psychiatric barriers that preclude understanding of informed consent process.
2. Patients in which the site investigator is unable to comply with completion of study documentation following PCI, i.e. patients with planned transfer to another hospital not participating in the registry.
3. Enrollment in a clinical trial involving another anticoagulant agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UA, STEMI and NSTEMI ACS patients treated prior to PCI with LMWH and/or patients treated with LMWH during PCI i.e. in catheterization laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 747 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Description of anticoagulant management during PCI and current practices of participating centres will be undertaken | in-hospital

SECONDARY OUTCOMES:
In-hospital safety outcomes including - major, minor bleeding, requirement for transfusion, death, myocardial infarction (or re-MI), myocardial ischemia requiring urgent revascularization, and major bleeding | in-hospital
In-hospital angiographic complications: no reflow, thrombus, occlusion of collateral branches, distal embolism, coronary dissection, acute closure of the culprit vessel | in-hospital
PCI-related resources utilization during the study period, including cost of PCI and its treatment (e.g. duration of hospital stay, drug costs, costs related to bleeding such as transfusions) | in-hospital

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada